CLINICAL TRIAL: NCT03855189
Title: Safety and Efficacy of SCH 32088 vs Beclomethasone Dipropionate (Vancenase AQ) and Placebo in Seasonal Allergic Rhinitis
Brief Title: Safety and Efficacy of Mometasone Furoate (SCH 032088) vs Beclomethasone Dipropionate or Placebo in Seasonal Allergic Rhinitis (C93-013)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C93-013; C93-013 (Other: Merck)
Record Dates: First submitted 2019-02-25; First posted 2019-02-26 (Actual); Results first posted 2019-08-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mometasone Furoate (MF) (Experimental): Participants receive 200 mcg nasal MF in the morning upon awakening and placebo approximately 12 hours later in the evening (200 mcg total daily dose) for 29 days.
  Interventions: Drug: Mometasone Furoate (MF); Drug: Placebo
- Beclomethasone Dipropionate (BDP) (Active Comparator): Participants receive 168 mcg nasal BDP in the morning upon awakening and an additional 168 mcg approximately 12 hours later in the evening (336 mcg total daily dose) for 29 days.
  Interventions: Drug: Beclomethasone Dipropionate (BDP)
- Placebo (Placebo Comparator): Participants receive nasal placebo in the morning upon awakening and again approximately 12 hours later in the evening for 29 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone Furoate (MF) — Mometasone furoate nasal spray administered as 200 mcg total dose per day for 4 weeks.
  Other Names: SCH 032088; MK-0887; Nasonex®
  Arms: Mometasone Furoate (MF)
Drug: Beclomethasone Dipropionate (BDP) — Beclomethasone dipropionate nasal spray administered as 168 mcg twice daily (BID) [336 mcg total dose per day] for 4 weeks.
  Other Names: Vancenase® AQ
  Arms: Beclomethasone Dipropionate (BDP)
Drug: Placebo — Placebo nasal spray administered for 4 weeks.
  Arms: Mometasone Furoate (MF); Placebo

SUMMARY:
The objectives of this study are to determine the safety and efficacy in seasonal allergic rhinitis of a four-week course of mometasone furoate compared to beclomethasone dipropionate or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant women of childbearing potential must be using a medically acceptable form of birth control for at least 3 months prior to Screening, and must continue its use for the duration of the study. Women not of childbearing potential must be surgically sterilized or at least one year post menopausal, or be otherwise incapable of bearing children
* 2-year history of seasonal allergic rhinitis
* Positive skin test response to a local seasonal allergen within last 2 years
* Good health and free of any unstable, clinically significant disease, other than allergic rhinitis, that would interfere with the study schedule or evaluation of seasonal allergic rhinitis

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Women of childbearing potential who are not using an acceptable form of birth control
* Pre-menarchal females
* Asthma requiring therapy with inhaled or systemic corticosteroids
* Significant renal, hepatic, neurologic, cardiovascular, hematologic, metabolic, cerebrovascular, respiratory, gastrointestinal, or other significant medical illness or disorder which, in the judgment of the investigator, may interfere with the study, or require treatment which might interfere with the study
* On immunotherapy (unless maintenance therapy)
* Upper respiratory tract or sinus infection that requires antibiotic therapy within the previous 2 weeks
* Use of any investigational drug within the previous 90 days unless the investigational drug is a nasal corticosteroid or has a short (12 hours or less) duration of action, in which case the washout period will be 30 days
* Large nasal polyps, marked septal deviations or any other nasal structural abnormality that significantly interferes with nasal air flow
* Allergy to corticosteroids, or a history of multiple drug allergies
* History of posterior subcapsular cataracts
* Dependence upon nasal, oral or ocular decongestants or who are diagnosed with rhinitis medicamentosa
* Chronic use of any medication which could affect the course of seasonal allergic rhinitis
* Clinically significant abnormal electrocardiogram (ECG)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 1993-08-23 (Actual); Primary Completion 1993-10-08 (Actual); Study Completion 1993-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate (MF): Participants received 200 mcg nasal MF in the morning upon awakening and placebo approximately 12 hours later in the evening (200 mcg total daily dose) for 29 days.
- Beclomethasone Dipropionate (BDP): Participants received 168 mcg nasal BDP in the morning upon awakening and an additional 168 mcg approximately 12 hours later in the evening (336 mcg total daily dose) for 29 days.
- Placebo: Participants received nasal placebo in the morning upon awakening and again approximately 12 hours later in the evening for 29 days.
Period: Overall Study
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Started | 113 | 116 | 116
Treated | 112 (Does not include 1 participant who received first dose but was excluded from safety analysis.) | 116 | 116
Completed | 103 | 109 | 110
Not Completed | 10 | 7 | 6
Not completed — Adverse Event | 5 | 2 | 4
Not completed — Treatment Failure | 1 | 1 | 2
Not completed — Noncompliance with Protocol | 0 | 1 | 0
Not completed — Did Not Return | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo | Total
Number analyzed (Participants) | 113 | 116 | 116 | 345
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (12.3) | 34.6 (12.1) | 35.5 (11.2) | 34.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 52 | 72 | 176
  Male | 61 | 64 | 44 | 169

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Total Nasal Symptom Score (TNSS) (Average of Morning [AM]/Evening [PM] Score) Averaged Over Days 1 to 15 (Participant-Evaluated)
Description: TNSS evaluated participant nasal symptoms of discharge (rhinorrhea), stuffiness, sneezing, and itching, as rated in their diary in the morning (AM) and evening (PM). The 4 individual symptom scores rated as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe. TNSS was the sum of the 4 individual symptom scores (range= 0-12, higher score indicating more frequent/severe nasal symptoms). For the 15 day interval, participant individual daily scores were totaled and averaged over interval (AM and PM computed separately then averaged) and used to calculate the overall average change from Baseline. Participant average changes were then used to calculate the mean change for each arm for the interval. Average change from Baseline for Days 1-15 = average post-treatment score (Days 1-15) - Baseline average score (average of the Baseline AM/PM diary scores from 3 consecutive days prior to Baseline visit). Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline, and Days 1 through 15 (average of 15 days of treatment)
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available diary data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
score on a scale
  Baseline | 7.6 (2.2) | 7.3 (2.2) | 7.6 (2.0)
  Change from Baseline Days 1-15 | -2.3 (2.7) | -2.8 (2.1) | -1.5 (2.1)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from ANOVA; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from ANOVA; Test type: Other; p = 0.06, ANOVA

2. Secondary Outcome: Change From Baseline in the TNSS At Day 4 (Physician-Evaluated)
Description: TNSS evaluated participant nasal symptoms of discharge (rhinorrhea), stuffiness, sneezing, and itching. The 4 individual symptom scores were rated by the physician at the visit as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe. TNSS was the sum of the 4 individual symptom scores (range= 0-12, higher score indicating more frequent/severe nasal symptoms). For each participant, individual scores were totaled and used to calculate the change from Baseline in TNSS at the visit. Participant changes were then used to calculate the mean change for each treatment group at that visit. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1), Day 4
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 4 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 8.3 (1.7) | 7.9 (1.7) | 8.4 (1.6)
  Change From Baseline Day 4: number analyzed (Participants) | 110 | 113 | 116
  Change From Baseline Day 4 | -2.4 (2.8) | -2.7 (2.2) | -1.8 (2.5)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.04, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.50, ANOVA

3. Primary Outcome: Number of Participants Who Experienced ≥1 Adverse Event
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants with at least one AE was reported for each treatment group.
Time Frame: Up to 31 Days
Population: All randomized participants who received at least one dose of study medication and had at least one post-Baseline evaluation were analyzed for safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 112 | 116 | 116
Participants | 60 | 64 | 78

4. Primary Outcome: Number of Participants Who Discontinued Treatment Due to An Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants who discontinued due to an AE was reported for each treatment group.
Time Frame: Up to 31 Days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 112 | 116 | 116
Participants | 5 | 2 | 4

5. Secondary Outcome: Change From Baseline in the TNSS At Day 8 (Physician-Evaluated)
Description: as for outcome 2
Time Frame: Baseline (Day 1), Day 8
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 8 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 8.3 (1.7) | 7.9 (1.7) | 8.4 (1.6)
  Change From Baseline Day 8: number analyzed (Participants) | 110 | 113 | 113
  Change From Baseline Day 8 | -3.3 (2.9) | -3.8 (2.3) | -1.9 (2.7)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.11, ANOVA

6. Secondary Outcome: Change From Baseline in the TNSS At Day 15 (Physician-Evaluated)
Description: as for outcome 2
Time Frame: Baseline (Day 1), Day 15
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 15 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 8.3 (1.7) | 7.9 (1.7) | 8.4 (1.6)
  Change From Baseline Day 15: number analyzed (Participants) | 107 | 111 | 112
  Change From Baseline Day 15 | -3.3 (2.9) | -3.8 (2.7) | -2.6 (2.5)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.05, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.13, ANOVA

7. Secondary Outcome: Change From Baseline in the TNSS At Day 22 (Physician-Evaluated)
Description: as for outcome 2
Time Frame: Baseline (Day 1), Day 22
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 22 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 8.3 (1.7) | 7.9 (1.7) | 8.4 (1.6)
  Change From Baseline Day 22: number analyzed (Participants) | 105 | 110 | 109
  Change From Baseline Day 22 | -3.9 (2.9) | -4.0 (2.7) | -3.2 (2.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.06, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.03, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.81, ANOVA

8. Secondary Outcome: Change From Baseline in the TNSS At Day 29 (Physician-Evaluated)
Description: as for outcome 2
Time Frame: Baseline (Day 1), Day 29
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 29 visit data for TNSS.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 8.3 (1.7) | 7.9 (1.7) | 8.4 (1.6)
  Change From Baseline Day 29: number analyzed (Participants) | 100 | 105 | 105
  Change From Baseline Day 29 | -4.1 (2.9) | -4.6 (2.6) | -3.2 (2.7)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.02, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.17, ANOVA

9. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 4 (Physician-Evaluated)
Description: Overall condition of seasonal allergic rhinitis was evaluated by the physician during the visit and scored on a scale from 0 to 3 as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe. A higher score indicated more frequent/severe nasal symptoms. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1), Day 4
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 4 visit data for SAR overall condition (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.3 (0.5) | 2.2 (0.4) | 2.2 (0.1)
  Change From Baseline Day 4: number analyzed (Participants) | 110 | 113 | 116
  Change From Baseline Day 4 | -0.6 (0.7) | -0.5 (0.7) | -0.3 (0.7)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.02, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.39, ANOVA

10. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 8 (Physician-Evaluated)
Description: as for outcome 9
Time Frame: Baseline (Day 1), Day 8
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 8 visit data for SAR overall condition (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.3 (0.5) | 2.2 (0.4) | 2.2 (0.1)
  Change From Baseline Day 8: number analyzed (Participants) | 110 | 113 | 113
  Change From Baseline Day 8 | -0.7 (0.8) | -0.8 (0.7) | -0.3 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.60, ANOVA

11. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 15 (Physician-Evaluated)
Description: as for outcome 9
Time Frame: Baseline (Day 1), Day 15
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 15 visit data for SAR overall condition (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.3 (0.5) | 2.2 (0.4) | 2.2 (0.1)
  Change From Baseline Day 15: number analyzed (Participants) | 107 | 111 | 112
  Change From Baseline Day 15 | -0.7 (0.8) | -0.8 (0.7) | -0.5 (0.7)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.03, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.54, ANOVA

12. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 22 (Physician-Evaluated)
Description: as for outcome 9
Time Frame: Baseline (Day 1), Day 22
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 22 visit data for SAR overall condition (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.3 (0.5) | 2.2 (0.4) | 2.2 (0.1)
  Change From Baseline Day 22: number analyzed (Participants) | 105 | 110 | 109
  Change From Baseline Day 22 | -0.9 (0.8) | -0.8 (0.7) | -0.6 (0.7)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.71, ANOVA

13. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 29 (Physician-Evaluated)
Description: as for outcome 9
Time Frame: Baseline (Day 1), Day 29
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 29 visit data for SAR overall condition (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.3 (0.5) | 2.2 (0.4) | 2.2 (0.1)
  Change From Baseline Day 29: number analyzed (Participants) | 100 | 105 | 105
  Change From Baseline Day 29 | -0.9 (0.9) | -0.9 (0.8) | -0.6 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.77, ANOVA

14. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 4 (Participant-Evaluated)
Description: Overall condition of seasonal allergic rhinitis was evaluated by the participant during the visit and scored on a scale from 0 to 3 as follows: 0 = none, 1 = mild, 2 = moderate, 3 = severe. A higher score indicated more frequent/severe nasal symptoms. Change from Baseline = visit score - Baseline score (Day 1 visit). Negative changes from baseline indicate a decrease in symptom severity.
Time Frame: Baseline (Day 1), Day 4
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 4 visit data for SAR overall condition (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.2 (0.5) | 2.2 (0.5) | 2.3 (0.5)
  Change From Baseline Day 4: number analyzed (Participants) | 110 | 113 | 116
  Change From Baseline Day 4 | -0.6 (0.8) | -0.6 (0.6) | -0.4 (0.7)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.11, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.03, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.60, ANOVA

15. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 8 (Participant-Evaluated)
Description: as for outcome 14
Time Frame: Baseline (Day 1), Day 8
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 8 visit data for SAR overall condition (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.2 (0.5) | 2.2 (0.5) | 2.3 (0.5)
  Change From Baseline Day 8: number analyzed (Participants) | 110 | 113 | 112
  Change From Baseline Day 8 | -0.7 (0.8) | -0.8 (0.7) | -0.4 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.59, ANOVA

16. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 15 (Participant-Evaluated)
Description: as for outcome 14
Time Frame: Baseline (Day 1), Day 15
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 15 visit data for SAR overall condition (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.2 (0.5) | 2.2 (0.5) | 2.3 (0.5)
  Change From Baseline Day 15: number analyzed (Participants) | 107 | 111 | 112
  Change From Baseline Day 15 | -0.7 (0.8) | -0.8 (0.8) | -0.5 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.07, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.43, ANOVA

17. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 22 (Participant-Evaluated)
Description: as for outcome 14
Time Frame: Baseline (Day 1), Day 22
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 22 visit data for SAR overall condition (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.2 (0.5) | 2.2 (0.5) | 2.3 (0.5)
  Change From Baseline Day 22: number analyzed (Participants) | 105 | 110 | 109
  Change From Baseline Day 22 | -0.9 (0.8) | -0.9 (0.8) | -0.7 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.09, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.08, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.96, ANOVA

18. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis At Day 29 (Participant-Evaluated)
Description: as for outcome 14
Time Frame: Baseline (Day 1), Day 29
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 29 visit data for SAR overall condition (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 111 | 113 | 116
scores on a scale
  Baseline | 2.2 (0.5) | 2.2 (0.5) | 2.3 (0.5)
  Change From Baseline Day 29: number analyzed (Participants) | 100 | 105 | 104
  Change From Baseline Day 29 | -0.9 (0.9) | -0.9 (0.7) | -0.6 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.64, ANOVA

19. Secondary Outcome: Response To Therapy At Day 4 (Physician-Evaluated)
Description: Response to therapy was evaluated by the physician and based upon the participant's status scored relative to Baseline. Response was scored on a scale from 1 to 5 as follows: 1 = Complete Relief, 2 = Marked Relief, 3 = Moderate Relief, 4= Slight Relief, and 5 = Treatment Failure. A higher score indicated a weaker response.
Time Frame: Day 4
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 4 visit data for response (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 110 | 113 | 116
scores on a scale | 3.3 (1.2) | 3.2 (1.1) | 3.5 (1.1)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.25, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.02, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.26, ANOVA

20. Secondary Outcome: Response To Therapy At Day 8 (Physician-Evaluated)
Description: as for outcome 19
Time Frame: Day 8
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 8 visit data for response (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 110 | 113 | 113
scores on a scale | 3.0 (1.2) | 2.7 (1.1) | 3.5 (1.1)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.09, ANOVA

21. Secondary Outcome: Response To Therapy At Day 15 (Physician-Evaluated)
Description: as for outcome 19
Time Frame: Day 15
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 15 visit data for response (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 107 | 111 | 112
scores on a scale | 3.0 (1.1) | 2.8 (1.0) | 3.3 (1.0)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.05, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.07, ANOVA

22. Secondary Outcome: Response To Therapy At Day 22 (Physician-Evaluated)
Description: as for outcome 19
Time Frame: Day 22
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 22 visit data for response (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 105 | 110 | 109
scores on a scale | 2.8 (1.1) | 2.7 (1.1) | 3.1 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.04, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.53, ANOVA

23. Secondary Outcome: Response To Therapy At Day 29 (Physician-Evaluated)
Description: as for outcome 19
Time Frame: Day 29
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 29 visit data for response (physician-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 100 | 105 | 105
scores on a scale | 2.9 (1.2) | 2.5 (1.2) | 3.2 (1.2)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.02, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.02, ANOVA

24. Secondary Outcome: Response To Therapy At Day 4 (Participant-Evaluated)
Description: Response to therapy was evaluated by the participant and based upon their status scored relative to Baseline. Response was scored on a scale from 1 to 5 as follows: 1 = Complete Relief, 2 = Marked Relief, 3 = Moderate Relief, 4= Slight Relief, and 5 = Treatment Failure. A higher score indicated a weaker response.
Time Frame: Day 4
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 4 visit data for response (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 110 | 113 | 116
scores on a scale | 3.3 (1.0) | 3.2 (0.9) | 3.6 (0.9)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.03, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.34, ANOVA

25. Secondary Outcome: Response To Therapy At Day 8 (Participant-Evaluated)
Description: as for outcome 24
Time Frame: Day 8
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 8 visit data for response (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 110 | 113 | 113
scores on a scale | 3.0 (1.0) | 2.7 (1.0) | 3.5 (1.0)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.04, ANOVA

26. Secondary Outcome: Response To Therapy At Day 15 (Participant-Evaluated)
Description: as for outcome 24
Time Frame: Day 15
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 15 visit data for response (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 107 | 111 | 112
scores on a scale | 3.0 (1.1) | 2.7 (0.9) | 3.3 (1.0)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.06, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.03, ANOVA

27. Secondary Outcome: Response To Therapy At Day 22 (Participant-Evaluated)
Description: as for outcome 24
Time Frame: Day 22
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 22 visit data for response (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 105 | 110 | 109
scores on a scale | 2.9 (1.1) | 2.7 (1.1) | 3.1 (1.1)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.13, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.07, ANOVA

28. Secondary Outcome: Response To Therapy At Day 29 (Participant-Evaluated)
Description: as for outcome 24
Time Frame: Day 29
Population: All randomized participants who met eligibility criteria and evaluability criteria, completed at least one valid post-Baseline visit, and had available Day 29 visit data for response (participant-evaluated).
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
Number analyzed (Participants) | 100 | 105 | 104
scores on a scale | 2.9 (1.1) | 2.6 (1.1) | 3.3 (1.1)
Statistical Analysis 1: Comparison: Mometasone Furoate (MF) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.03, ANOVA
Statistical Analysis 2: Comparison: Beclomethasone Dipropionate (BDP) vs Placebo; Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate (MF) vs Beclomethasone Dipropionate (BDP); Pairwise treatment comparison based on t-test from an analysis of variance (ANOVA); Test type: Other; p = 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 31 Days
Description: All randomized participants who received at least one dose of study medication and had at least one post-Baseline evaluation were analyzed for safety.
Arm/Group | Mometasone Furoate (MF) | Beclomethasone Dipropionate (BDP) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/116 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 47/112 | 38/116 | 53/116
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate (MF) (N=112) | Beclomethasone Dipropionate (BDP) (N=116) | Placebo (N=116)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 3 (6) | 6 (13)
HEADACHE (Nervous system disorders) | 29 (59) | 27 (49) | 30 (66)
SINUS HEADACHE (Nervous system disorders) | 11 (14) | 6 (8) | 6 (10)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 6 (15) | 12 (28)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 6 (11) | 6 (9)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 8 (23)

LIMITATIONS AND CAVEATS:
AE Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 12.0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 30 days prior to submission for publication or presentation to review copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the Protocol study. Sponsor shall have editorial rights with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to proprietary information and the accuracy of the information contained in the publication.